CLINICAL TRIAL: NCT06097663
Title: A Randomized, Placebo-controlled, Parallel-group, Investigator- and Participant-blinded Phase 2a Study to Investigate the Efficacy, Safety, and Tolerability of DFV890 and MAS825 for Inflammatory Marker Reduction in an Adult Population With Coronary Heart Disease and Clonal Hematopoiesis of Indeterminate Potential (CHIP)
Brief Title: A Study to Investigate the Efficacy, Safety, and Tolerability of DFV890 and MAS825 for Inflammatory Marker Reduction in Adult Participants With Coronary Heart Disease and Clonal Hematopoiesis of Indeterminate Potential (CHIP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CADPT15A12201; 2023-506741-34-00 (Other: EU CTIS)
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Coronary Heart Disease; Clonal Hematopoiesis of Indeterminate Potential (CHIP)
Keywords: coronary heart disease; CHIP; inflammatory marker reduction; NLRP3 inflammasome inhibitor
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment Sequence 1 (Experimental): Treatment Sequence 1
  Interventions: Drug: MAS825; Drug: DFV890 placebo
- Treatment Sequence 2 (Experimental): Treatment Sequence 2
  Interventions: Drug: MAS825 Placebo; Drug: DFV890; Drug: DFV890 placebo
- Treatment Sequence 3 (Experimental): Treatment Sequence 3
  Interventions: Drug: MAS825 Placebo; Drug: DFV890; Drug: DFV890 placebo
- Treatment Sequence 4 (Experimental): Treatment Sequence 4
  Interventions: Drug: MAS825 Placebo; Drug: DFV890
- Treatment Sequence 5 (Placebo Comparator): Treatment Sequence 5
  Interventions: Drug: MAS825 Placebo; Drug: DFV890 placebo

INTERVENTIONS:
Drug: MAS825 — Active MAS825 single dose
  Arms: Treatment Sequence 1
Drug: MAS825 Placebo — MAS825 placebo single dose
  Arms: Treatment Sequence 2; Treatment Sequence 3; Treatment Sequence 4; Treatment Sequence 5
Drug: DFV890 — Oral tablet of DFV890 active once daily
  Arms: Treatment Sequence 2; Treatment Sequence 3; Treatment Sequence 4
Drug: DFV890 placebo — Oral tablet of DFV890 placebo once daily
  Arms: Treatment Sequence 1; Treatment Sequence 2; Treatment Sequence 3; Treatment Sequence 5

SUMMARY:
This Phase 2a clinical trial will evaluate the effectiveness, safety, and tolerability of increasing dose strengths of an oral daily medication, DFV890, administered for 12 weeks, or a single s.c. dose of MAS825, to reduce key markers of inflammation related to CVD risk, such as IL-6 and IL-18, in approximately 28 people with known coronary heart disease and TET2 or DNMT3A CHIP (VAF ≥2%).

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo-controlled, participant- and investigator-blinded study.

The study consists of a screening period up to 30 days; a treatment period of approximately 12 weeks with an end of treatment (EOT) visit on Day 85, which is one day after the last dose of DFV890 or placebo; a follow-up period of approximately 1 week; and a standard safety follow-up call approximately 30 days following the last dose. The overall study duration is approximately 21 weeks.

Participants will be randomized to one of five treatment sequences. Based on the treatment sequence assignments, participants will start on either a combination of MAS825 and placebo, DFV890 and placebo, or placebo and placebo on Day 1, and then, within each DFV890 treatment sequence, participants will receive up-titrating doses of DFV890 or placebo at the corresponding study visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged between 18 - 80 years (inclusive) at the start of screening will be included.
* Participants must have a body mass index (BMI) within the range of 18 - 40 kg/m2 at screening. BMI = Body weight (kg) / [Height (m)]2.
* Documented spontaneous myocardial infarction (MI) (diagnosed according to the universal MI criteria with or without evidence of ST segment elevation) at least 30 days before the start of screening (Thygesen et al 2007).
* Known presence of CHIP, restricted to driver mutations in TET2 or DNMT3A with a VAF ≥2%, as documented in the participant's medical history.
* For participants on statin therapy (HMG-CoA reductase inhibitor) as clinically indicated, participants must be on a stable regimen (at least 4 weeks before randomization), with no planned statin dose changes over the course of the trial treatment period. Unplanned statin dose changes during the trial treatment period may occur.

Exclusion Criteria:

* Patients receiving concomitant medications that are known to be strong or moderate inducers of cytochrome CYP2C9 enzyme and/or strong inducers of CYP3A, strong inhibitors of CYP2C9 and/or strong or moderate inhibitors of CYP3A and the treatment cannot be discontinued or switched to a different medication within 5 half-lives or 1 week (whichever is longer) prior to Day 1 and for the duration of the study.
* At screening, pre-malignant clonal cytopenias or clonal cytopenia of unknown significance (CCUS).
* History of ongoing, chronic, or major recurrent infectious disease, at the discretion of the Investigator, at the start of screening.
* Patients with suspected or proven immunocompromised state at screening.
* Use of any biologic drugs targeting the immune system within 26 weeks of Day 1.
* Multi-vessel coronary artery bypass graft (CABG) surgery within the past 3 years prior to the start of screening.
* Planned coronary revascularization (percutaneous coronary intervention (PCI) or CABG) or any other major surgical procedure during the study (until End of Study (EOS)).
* Symptomatic Class IV heart failure (New York Heart Association [NYHA]) at the start of screening.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Serum levels of IL-6 and IL-18 | From Day 22 to Day 92 (end of study)
  To evaluate the effect of various dose levels of DFV890 versus placebo to reduce circulating levels of inflammatory markers in participants with coronary heart disease and CHIP
Serum level of IL-6 | Day 22
  To evaluate the effect of MAS825 versus placebo to reduce circulating levels of inflammatory markers in participants with coronary heart disease and CHIP.

SECONDARY OUTCOMES:
Plasma trough concentrations (Ctrough) of DFV890 at steady-state | From Day 22 to Day 92
  To assess the pharmacokinetics of DFV890 in participants with coronary heart disease and CHIP.
Serum concentrations of MAS825 after a single s.c. dose of MAS825 | From Day 1 to Day 85
  To assess the pharmacokinetics of MAS825 in participants with coronary heart disease and CHIP.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (2):
  - Washington University, St Louis, Missouri
  - Vanderbilt University Medical Cent, Nashville, Tennessee
- Novartis Investigative Site, Montreal, Quebec, Canada
- Germany (3):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, München

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sumida K, Obeng EA, Kovesdy CP. Clonal Hematopoiesis in Kidney Disease. Clin J Am Soc Nephrol. 2025 Sep 11. doi: 10.2215/CJN.0000000895. Online ahead of print. No abstract available. PMID 40932796